CLINICAL TRIAL: NCT06178289
Title: The Effectiveness of 3M Cavilon Advanced Skin Protectant in the Treatment of Partial-thickness Wounds Caused by Moisture-associated Skin Damage Compared to Usual Wound Care Treatment in Hospitals: a Multi-centre RCT
Brief Title: Effectiveness of 3M Cavilon Advanced Skin Protectant in the Treatment of Moisture-associated Skin Damage in Hospitals
Acronym: ISR-CASP-MASD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2022-0527
Record Dates: First submitted 2023-11-30; First posted 2023-12-20 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Irritant Dermatitis; Stoma Site Dermatitis; Wound of Skin
MeSH Terms: conditions — Dermatitis, Irritant

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single: Investigator (central assessor of the photographs) will be blinded.
  The participants and care providers cannot be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 3M Cavilon Advanced Skin Protectant (Experimental): 3M Cavilon Advanced Skin Protectant (2,7ml) is a cyanoacrylate based film and will be administered every third day for a study period of 21 days.
  Interventions: Device: 3M Cavilon Advanced Skin Protectant
- Standard hospital wound treatment protocol (Active Comparator): Usual wound treatment care provided in the hospital will be administered.
  Interventions: Device: Standard hospital wound treatment protocol

INTERVENTIONS:
Device: 3M Cavilon Advanced Skin Protectant — 3M Cavilon Advanced Skin Protectant is applied to the study area of partial-thickness wounds (IAD category 2A, peri-wound MASD, peri-stomal MASD). Application of the study device should be according to the manufacturer's IFU. Comprehensive training for nurses will be provided to the study nurses.
  Other Names: cyanoacrylate based film
  Arms: 3M Cavilon Advanced Skin Protectant
Device: Standard hospital wound treatment protocol — Comparator: Standard hospital wound treatment protocol
  Arms: Standard hospital wound treatment protocol

SUMMARY:
Objectives: The aim of this study is to evaluate the effectiveness of 3M™ Cavilon™ Advanced Skin Protectant in the treatment of partial-thickness wounds caused by moisture (MASD) compared to usual wound care treatment.

Methodology:

RESEARCH DESIGN: A randomized controlled multicentre clinical trial.

DATA COLLECTION:

Randomization/Blinding and Participant Numbering: The patients will be allocated 1:1 by block randomization, using the REDCap Randomization Module, to either Cavilon™ Advanced Skin Protectant or local hospital partial-thickness wound (MASD) treatment protocol, yielding one study group. Due to the obvious differences between the comparative hospital wound care treatment products and the study device, the study nurses cannot be blinded. A blinded assessor will centrally assess the time to healing and other healing outcomes based on the photographs of the study area.

Study area: Defined as all partial-thickness, skin damaged areas on the body - due to exposure to (a) incontinence body fluids, (b) wound exudate, (c) stomal- or fistula effluent or digestive secretions.

Study duration: 21 days or until complete healing of the moisture associated skin damage (complete epithelialization).

Skin (MASD) assessment: Daily skin assessment of the study area is to be conducted by the study nurses. Relevant wound and patient information will be recorded (incontinence status, presence of a urinary catheter or faecal management system, number of absorbent pad or diaper changes, number of cleansing procedures, type of stoma, number of applications regarding Cavilon Advanced Skin Protectant or usual hospital wound treatment protocol). Digital planimetry software (PictZar® version 7.6.1 ss) will be the main mode of assessing wound healing. Therefore, daily photographs will be taken with each daily skin assessment after removal of all visual product to ensure blinded skin assessment by the central reviewer.

Pain assessment: The Numeric Rating Scale (NRS) or Crital care Pain Observation Tool (CPOT) will be used to assess pain daily. Treatment-related pain (pain experienced during treatment (cleansing and product application)) and wound related pain (pain perception specifically caused by the MASD lesion) will be assessed.

Nursing time assessment: Time per cleansing and time per treatment application.

DETAILED DESCRIPTION:
Problem statement:

Partial-thickness wounds (erosion/denudation of the epithelial and dermal layers of the skin) can occur due to prolonged exposure of moisture and irritants. Various sources of moisture can cause these superficial wounds called moisture-associated skin damage (MASD) which include wound exudate, bodily fluids from incontinence and effluent from stomas and fistulas. MASD can present as inflammation with or without erosion and even secondary infection. Partial-thickness denudation can be extremely painful and detrimental to the patient. Traditionally a wide array of treatment options is used in clinical practice, yet there is a lack of robust studies comparing newer technologies with current practices. 3M™ Cavilon™ Advanced Skin Protectant, launched in 2017, is a newer cyanoacrylate-based medical device indicated for treatment of partial-thickness skin loss and is the only cyanoacrylate-based barrier product available on the Belgian market.

Objectives: The aim of this study is to evaluate the effectiveness of 3M™ Cavilon™ Advanced Skin Protectant in the treatment of partial-thickness wounds caused by moisture (MASD) compared to usual wound care treatment.

Methodology:

RESEARCH DESIGN: A randomized controlled multicentre clinical trial.

DATA COLLECTION:

Procedure: Demographics and Participant Characteristics: Patient demographics will be recorded in REDCap eCRFs on study schedule Day 01: gender, age, height, weight, co-morbidities.

Randomization/Blinding and Participant Numbering: The patients will be allocated 1:1 by block randomization, using the REDCap Randomization Module, to either Cavilon™ Advanced Skin Protectant or local hospital partial-thickness wound (MASD) treatment protocol, yielding one study group. Due to the obvious differences between the comparative hospital wound care treatment products and the study device, the study nurses cannot be blinded. A blinded assessor will assess the time to healing and other healing outcomes centrally based on the photographs of the study area.

Study area: Defined as all partial-thickness, skin damaged areas on the body - due to exposure to (a) incontinence body fluids, (b) wound exudate, (c) stomal- or fistula effluent or digestive secretions.

Study duration: 21 days or until complete healing of the moisture associated skin damage (complete epithelialization).

Hypothesis: 3M™ Cavilon™ Advanced Skin Protectant is more effective in the treatment of partial-thickness wounds caused by moisture (moisture-associated skin damage) compared to usual wound care treatment in hospitals.

Skin (MASD) assessment: Daily skin assessment of the study area is to be conducted by the study nurses. Relevant wound and patient information will be recorded. This information includes incontinence status, presence of a urinary catheter or faecal management system, number of absorbent pad or diaper changes, number of cleansing procedures, type of stoma, number of applications regarding Cavilon Advanced Skin Protectant or usual hospital wound treatment protocol. Daily photographs will be taken with each daily skin assessment after removal of all visual product to ensure blinded skin assessment by the central reviewer. Digital planimetry software (PictZar® version 7.6.1 ss) will be the main mode of assessing wound healing. The central reader will perform a blinded skin assessment based on the provided photographic documentation of the study area.

Pain assessment: The Numeric Rating Scale (NRS) or Crital care Pain Observation Tool (CPOT) will be used to assess pain daily. Treatment-related pain (pain experienced during treatment (cleansing and product application)) and wound related pain (pain perception specifically caused by the MASD lesion) will be assessed.

Nursing time assessment: Time per cleansing and time per treatment application will be done on days 4 and 7 using a stopwatch.

DATA ANALYSIS:

All quantitative data will be summarized with descriptive statistics.

Inferential analysis: Cox proportional hazards will be used to calculate the primary efficacy variable. Linear mixed logistic regressions and linear mixed models will be used to calculate the secondary objectives.

Exploratory analysis: Cox proportional hazards will be used to calculate the primary efficacy variable. Linear mixed logistic regressions and linear mixed models will be used to calculate the secondary objectives.

Health economic evaluation: A cost-effectiveness analysis will be performed with an institutional perspective in a Belgian context. Total cost will be calculated by the sum of the total product cost and the total cost of nursing time. Costs will be averaged within each group and compared using a two-signed t-test at an alpha level of 5%. A cost-effectiveness analysis will be performed by calculating the ICER. The ICER will be expressed in euros per wound healed per patient.

ELIGIBILITY:
Inclusion Criteria:

* The patient or their legally authorized representative signed informed consent.
* The patient is expected to be in the study for the full duration of the trial.
* The patient has partial thickness wounds caused by moisture (MASD) i.e.,

  * The patient has IAD category 2A or
  * Peri-wound MASD or
  * Peri-stomal MASD.

Exclusion Criteria:

* Patients with a known hypersensitivity or allergy to acrylate or cyanoacrylate.
* The patient requires topical treatment due to a fungal, bacterial or viral infection in the study area.
* Intertriginous dermatitis (most often a fungal infection is present).
* Peri-fistula MASD (would usually require hospitalization).
* The patient has any other local dermatological disease or skin condition interfering with this study.
* Patients participating in another study with a known or implied effect on skin barrier function.
* Patients who are receiving end-of-life care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Time to complete epithelialization | Day 01 - Day 21
  Number of days from commencement of application of study device or comparator to the study area to complete resolution of partial-thickness wound

SECONDARY OUTCOMES:
Proportion of participants with complete epithelialization | Day 07, Day 14, Day 21
  The proportion of patients with partial-thickness wounds completely healed at days 7, 14 and 21
Mean change in treatment related pain | Day 01 - Day 21
  The mean change in patients' perception of treatment-related pain using the Wong-Baker FACES Pain Rating Scale from baseline to day 21.
Mean change in wound pain | Day 01, Day 02, Day 04, Day 07
  The mean change in patients' perception of wound pain using the Wong-Baker FACES Pain Rating Scale before treatment, 30 minutes after the first treatment, 24 hours after the first treatment, on day 4, and on day 7.
Change in maceration surface area | Day 07, Day 14, Day 21
  The percent of change in maceration (area) at days 7, 14, and 21.
Total treatment cost | Day 04, Day 07
  To investigate the total cost of treating partial-thickness wounds including number of applications, product costs and nursing time assessments to measure time per cleansing and time per treatment application on day 4 and 7 (by researcher).

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, PhD, Principal Investigator — University Ghent
Locations (3):
- Belgium (3):
  - Ziekenhuis Aan de Stroom (ZAS), Antwerp
  - Ghent University Hospital, Ghent
  - AZ Oudenaarde, Oudenaarde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woo KY, Beeckman D, Chakravarthy D. Management of Moisture-Associated Skin Damage: A Scoping Review. Adv Skin Wound Care. 2017 Nov;30(11):494-501. doi: 10.1097/01.ASW.0000525627.54569.da. PMID 29049257
- [Background] Gray M, Black JM, Baharestani MM, Bliss DZ, Colwell JC, Goldberg M, Kennedy-Evans KL, Logan S, Ratliff CR. Moisture-associated skin damage: overview and pathophysiology. J Wound Ostomy Continence Nurs. 2011 May-Jun;38(3):233-41. doi: 10.1097/WON.0b013e318215f798. PMID 21490547
- [Background] Beeckman D, Van den Bussche K, Alves P, Arnold Long MC, Beele H, Ciprandi G, Coyer F, de Groot T, De Meyer D, Deschepper E, Dunk AM, Fourie A, Garcia-Molina P, Gray M, Iblasi A, Jelnes R, Johansen E, Karadag A, Leblanc K, Kis Dadara Z, Meaume S, Pokorna A, Romanelli M, Ruppert S, Schoonhoven L, Smet S, Smith C, Steininger A, Stockmayr M, Van Damme N, Voegeli D, Van Hecke A, Verhaeghe S, Woo K, Kottner J. Towards an international language for incontinence-associated dermatitis (IAD): design and evaluation of psychometric properties of the Ghent Global IAD Categorization Tool (GLOBIAD) in 30 countries. Br J Dermatol. 2018 Jun;178(6):1331-1340. doi: 10.1111/bjd.16327. Epub 2018 Apr 19. PMID 29315488